CLINICAL TRIAL: NCT03697694
Title: Randomized, Parallel, Double-blind, Placebo Controlled, Study in Men to Assess the Influence of Aronox on Parameters Associated With Aerobic Performance
Brief Title: To Assess the Influence of Aronox on Parameters Associated With Aerobic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Naturex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NUAR02
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2018-10

CONDITIONS: Aerobic Capacity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500mg of Aronox® >40% polyphenol aronia extract (Experimental): Name: Aronia PE 40% polyphenols Description: Powdered extract obtained from aronia berries (Aronia melanocarpa) Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg aronia extract Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX / Virage sante
  Interventions: Dietary Supplement: 500mg of Aronox® >40% polyphenol aronia extract
- 500mg of placebo (Placebo Comparator): Name: Placebo Description: Identical formulation as the treatment consisting of colored maltodextrin using artificial colors Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg placebo Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX (Advance nutraceutical) / Virage sante
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 500mg of Aronox® >40% polyphenol aronia extract — Name: Aronia PE 40% polyphenols Description: Powdered extract obtained from aronia berries (Aronia melanocarpa) Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg aronia extract Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX / Virage sante
  Arms: 500mg of Aronox® >40% polyphenol aronia extract
Other: Placebo — Name: Placebo Description: Identical formulation as the treatment consisting of colored maltodextrin using artificial colors Dosage form: Capsule (opaque, beige, size 00) Strength: 500 mg placebo Regimen 1 capsule, once a day with breakfast (except on days when attending the laboratory) Batch number: As per label Expiry Date: As per label Manufacturer: NATUREX (Advance nutraceutical) / Virage sante
  Arms: 500mg of placebo

SUMMARY:
A randomized, double blind, counterbalanced, placebo controlled independent groups design. Participants will then be familiarized with the ergometer to determine settings and seating position and randomized to an investigational product group (2 groups: Aronox vs placebo; 1:1 allocation). A time to undergo baseline testing will then be scheduled (day 0). On the baseline day, stature, body mass, blood pressure and heart rate will be assessed. Participants will then complete a submaximal aerobic performance test (lactate profile) where expired gas, heart rate, blood lactate,and RPE will be measured. Following a 10-min rest, participants will then perform a ramp test to exhaustion to determine VO2max (this will be to finalize eligibility to the study - VO2max of 45-70 ml/kg/min). Expired gas, heart rate, power output, perceived exertion, and near-infra-red spectroscopy will be collected throughout and blood lactate will be determined at test termination. Those that do not fulfill the criteria for VO2max will be excluded from the study at this point. Those that are eligible (verified by their VO2max) will consume a standardized 'light' meal and rest for 2 h. Time to exhaustion (TTE) trial (60%GET) determined from previous tests (lactate profile and VO2max) will then be completed. On completion of the TTE trial, the first dose of the investigational product will be administered in the laboratory and participants will be given a 4-week supply of the investigational product to take in the morning with breakfast. Participants will also be given study diaries to complete (exercise, general health, dietary intake). On the final study day (day 28), remaining investigational capsules and study diaries will be collected to monitor compliance. An identical trial to day 0 will then be conducted, following which participants will be asked if they knew what supplement they were asked to consume and be given the chance to provide feedback on their experience.

DETAILED DESCRIPTION:
Prior to the visit, participants will be issued with a participant information sheet to inform of the procedure and study requirements,then undergo initial screening via email or telephone to ascertain suitability to participate. If interested parties wish to participate, then an invitation for a familiarisation visit will be made, where they will:

Be provided with an overview of the protocol and given the opportunity to ask questions Complete a health and physical activity questionnaire to ascertain study suitability Complete a training status questionnaire Assessment of ability to swallow capsules Complete an informed consent to participate in the study (assuming they meet the criteria and are willing to participate)

Exercise protocol details During the first and second visit to the laboratory, participants will complete cycling tests; a submaximal exercise test and an incremental ramp exercise test to exhaustion to elucidate maximal aerobic power (Wmax), VO2max and gas exchange threshold (GET); both tests will be completed using an electro-magnetically braked cycle ergometer. The submaximal test will require participants to begin cycling at 100 W, which will increase by 25 W every minutes. Heart rate and capillary blood samples will taken from the earlobe in the last 30 s of each stage and immediately analysed for blood lactate concentration. Cycling will be terminated when the lactate turn-point had been reached. Throughout the submaximal test, near-infra-red spectroscopy (NIRS) and pulmonary gas exchange will be monitored through an online gas analysis system. Gas data will be averaged over the final 30 s of each stage in order to analyse the O2 cost. Following the completion of the submaximal test, participants will be given 10 minutes rest prior to completing the incremental ramp test to exhaustion to determine VO2max. The ramp test will consisted of 3 minutes of cycling at 100 W, followed by an increase in work rate of 1 W every 3 seconds (20 W.min-1) until the participant reaches volitional exhaustion or the cadence drops 10 rpm below the preferred cadence. Breath-by-breath pulmonary gas exchange data will collected throughout the ramp protocol and VO2max will be calculated as the highest 30-second average in oxygen consumption. Using the regression equation calculated from the submaximal VO2 data and the VO2max, it will then possible to identify the power output associated with the GET. The GET will be determined using either the first disproportionate increase in CO2 production (VCO2) from visual inspection of individual plots of VCO2 vs. VO2 or an increase in expired ventilatory equivalents (VE/VO2 with no increase in VE/VCO2). Following a standardized meal during a rest period of ~2 h, a time to exhaustion (TTE) test will be completed to examine exercise tolerance. The intensity for TTE test will be 60% of the difference between GET and VO2max. Saddle, handlebar height and fore/aft position was recorded and replicated on the return laboratory visit following supplementation.

Standardized meal Descriptive measures and a Physical Activity Level (PAL) of 1.7 will be used to calculate the participant's individual resting energy expenditure. This will subsequently identify the amount of cereal (Rice Snaps, Tesco, Manchester, UK) and semi-skimmed milk (1g/kg/bm) each individual will need to consume to meet 10% of their daily energy requirements (DER). This standardized fixed-energy breakfast meal will consist of a cereal: milk ratio of 30 g: 120 mL and will deliver fat, protein and carbohydrate with a macronutrient composition of 14, 14 & 72%, respectively.

Supplementation Following group allocation, participants will be provided with aronia (Aronox®) or placebo (PLA) supplementation and instructed to consume 500mg of the investigational product with breakfast every day for 4 weeks.

Data Analysis:

Statistical analysis will be performed using PASW Statistics 21.0 for Windows (SPSS, Inc., Chicago, IL.). All group characteristics will be reported as means ± standard errors, unless otherwise stated. A two-way ANOVA tests will be used to allow for comparison of between- and within- group mean differences for each dependent variable. Appropriate post-hoc analysis will be performed to determine any location of significance. Mauchley's test will

ELIGIBILITY:
Inclusion Criteria:

* Healthy men 18-50 years of age
* Not taking dietary supplement or pre workout supplements for at least 1 month prior to study start
* Perform between 4 and 20 hours of cycling per week
* VO2 max range ≥45 and <70 ml/kg/min
* Willing to participate and adhere to the study protocol
* Willing to not change their dietary / workout habits throughout the study
* Willing to limit berry and/or cherry intake to one portion per day
* Able to understand the participant information, health screening questionnaire and informed consent information
* Willing to participate and sign the informed consent form

Exclusion Criteria:

* BMI >30
* History or current cardiometabolic, gastrointestinal or renal diseases
* Taking any medication that might affect the outcome of the study, such as anti-inflammatory and immunosuppressant drugs.
* Performance enhancing drugs and recreational drugs
* Orthopedic problems that include muscle tears that might affect ability to perform exercise
* Have a recent history of surgery that might affect physical performance
* Smoking
* Recent or planned change in dietary habit
* Have lost more than 6 kg in the past 6 months or planning to lose weight in the next month
* Allergy to berries
* Drinking more than 2 alcoholic beverages per day on average in a week (total 14 units)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 59 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Change in time to fatigue | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox® on performance (time to fatigue) during high intensity cycling exercise (time to exhaustion trial) as compared to placebo

SECONDARY OUTCOMES:
VO2max | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox® vs Placebo on aerobic performance (respiratory gas analysis - V ̇O2max) during a ramp test to exhaustion
Blood lactate | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on markers of human performance (blood lactate) during a submaximal exercise test.

OTHER OUTCOMES:
Aerobic performance - submaximal test power output | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on power output during a submaximal exercise test
Aerobic performance - submaximal test heart rate | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on heart rate during a submaximal exercise test
Aerobic performance - submaximal test rate of perceived exertion | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on rate of perceived exertion during a submaximal exercise test
Aerobic performance- VO2max test power output | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance power output during an incremental ramp test until participant reaches volitional exhaustion during the VO2max test
Aerobic performance- VO2max test heart rate | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance heart rate during an incremental ramp test until participant reaches volitional exhaustion during the VO2max test
Aerobic performance- VO2max test rate of perceived exertion | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance rate of perceived exertion during an incremental ramp test until participant reaches volitional exhaustion during the VO2max test
Aerobic performance- time to exhaustion power output | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance power output during a time to exhaustion test
Aerobic performance- time to exhaustion blood lactate | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance blood lactate during a time to exhaustion test
Aerobic performance- time to exhaustion heart rate | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance heart rate during a time to exhaustion test
Aerobic performance- time to exhaustion rate of perceived exertion | Baseline and POST 28-35 day supplementation period
  Determine the effect of Aronox vs Placebo on other markers of aerobic performance rate of perceived exertion during a time to exhaustion test

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle, Tyne & Wear, United Kingdom